CLINICAL TRIAL: NCT04592601
Title: The S.L.I.M.M.S. Procedure for Severe Clinical Obesity
Acronym: SLIMMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The N.E.W. Program (Other)
Responsible Party: Principal Investigator, BRIAN B. QUEBBEMANN, M.D., F.A.C.S., Director, The N.E.W. Program
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLIMMS
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Morbid Obesity; Metabolic Syndrome; Type2 Diabetes; Insulin Resistance
Keywords: Obesity; Surgery; Bariatric Surgery; Morbid Obesity; Gastric Bypass; Sleeve Gastrectomy; SLIMMS
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Insulin Resistance; Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Prospective Single Group Clinical Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- S.L.I.M.M.S. Procedure (Experimental): Prospective collection of data on the safety and efficacy of the S.L.I.M.M.S. Procedure
  Interventions: Procedure: S.L.I.M.M.S. Procedure

INTERVENTIONS:
Procedure: S.L.I.M.M.S. Procedure — Combined Gastric Bypass with Vertical Sleeve Gastrectomy
  Other Names: Bariatric Surgery

SUMMARY:
Assessment of Gastric Bypass combined with Vertical Sleeve Gastrectomy as primary treatment for patients with severe clinical obesity.

Average percentage of total weight loss and percentage excess weight loss will be computed at 6 months, one year and then annually. Comorbid conditions, quality of life measures, appetite and satiety measures and adverse events will be tracked.

DETAILED DESCRIPTION:
BACKGROUND

Metabolic Disease and Obesity

Obesity is one of the most common chronic diseases in America and is strongly associated with additional metabolic disorders, in particular hypertension, dyslipidemia and insulin resistance. The combination of obesity with this cluster of metabolic disorders increases risk for cardiovascular disease and is widely recognized by the term Metabolic Syndrome.

According to the Centers for Disease Control, in 2017-2018 the "prevalence of severe obesity among U.S. adults was 9.2%", the "age-adjusted prevalence of obesity in adults was 42.4%", and the prevalence of metabolic syndrome (MS) in the obese population is higher than 60%. The economic impact of metabolic syndrome is significant, with risk factors for MS shown to increase a person's annual healthcare costs by more than $2000.

Efforts to treat obesity and obesity-associated metabolic disease currently include medical management and surgical intervention. Success rates with surgical interventions exceed those of medical management but are dependent on patients making permanent changes in eating behaviors.

Commonly accepted surgical procedures have several mechanisms of action. These include decreased stomach volume restricting a patient's ability to eat, intestinal bypass resulting in significant malabsorption, and alterations in hormonal control of appetite and satiety. Standardized surgical procedures include Vertical Sleeve Gastrectomy (VSG), Roux-en-Y Gastric Bypass (GBP), Laparoscopic Gastric Banding (LB) and Biliopancreatic Diversion with Duodenal Switch (DS). Of these, VSG and GBP are the most commonly performed.

VSG and GBP have been shown to result in similar weight loss, however, both procedures have a significant long-term failure rate.

Key symptomatic differences between VSG and GBP

During the initial 6-12 months after surgery, both VSG and GBP patients typically report a marked decrease in appetite as well as a significant restriction in volume of food that can be eaten before "feeling full." This period of decreased appetite and early satiety is commonly referred to as the "honeymoon period." After this honeymoon period, every patient's weight loss success becomes progressively more dependent on changes made in their eating habits.

As would be expected with anatomically distinct procedures, patient symptoms begin to significantly differ over time. Patients that have undergone GBP, resulting in a gastric pouch that is less than 30cc report a more sustained feeling of restriction in the volume of food that can be eaten at a single meal compared to patients that have undergone VSG with a 100-150cc residual stomach. GBP patients also report a more persistent feeling of early satiety than do patients after VSG. In contrast, patients that have undergone VSG, with most of the Ghrelin-producing region of their stomach removed, report a more persistent decrease in appetite compared to patients after GBP, where the production of Ghrelin appears to rebound.

Key hormonal differences between VSG and GBP

VSG results in substantial and permanent decrease in the orexigenic hormone Ghrelin. After GBP, rebound of Ghrelin is shown to occur within 6 to 12 months after surgery.

GBP causes a significantly greater increase in postprandial GLP-1 and Peptide YY, possibly contributing to earlier satiety and improved glycemic control.

Key differences in side effects between VSG and GBP

A common side effect of VSG is GERD. When symptoms are severe, conversion to GBP provides relief.

Dumping syndrome, a side effect of GBP, is often described as an effective negative feedback mechanism, helping to minimize ingestion of high glycemic index foods. Dumping is not typically associated with VSG.

Considering these differences, it is reasonable to question whether a single-stage procedure that combines the anatomic changes of both the GBP and VSG would result in;

1. Improved weight loss
2. An improved quality of life
3. Better glycemic control

PROPOSED STUDY

Surgical Intervention

The S.L.I.M.M.S. Procedure, for Surgically Limit Intake and Manage Metabolic Syndrome, is a single-stage operation combining Roux-en-Y Gastric Bypass with Partial Gastrectomy. The procedure specifications are listed below,

1. A 20 cc gastric pouch
2. A 10 mm diameter gastro-jejunal stoma
3. A 40 cm biliopancreatic limb (measured from the Ligament of Treitz)
4. A 150 cm roux limb
5. Resection of the remaining fundus and body of the stomach, maintaining the majority of the gastric antrum
6. Oversewing the gastric staple lines and buttressing with omentum

Most new procedures focus on variations of intestinal reconstruction, or involve implantation of artificial devices. The proposed procedure does not require implantation of an artificial device, nor a new method of intestinal reconstruction. It simply combines the two most common bariatric procedures in the world with the hope of providing cumulative benefits without increased risk.

Key Technical and Anatomic Precedents

1. When VSG results in severe and recalcitrant GERD the standard treatment is conversion to GBP. The final anatomic result is a patient with a gastric bypass and the majority of the gastric fundus and body removed. This is similar to the final anatomy of the procedure proposed in this study, however, the S.L.I.M.M.S. procedure will be done as a single operation.
2. In several centers, resectional gastric bypass, involving a standard gastric bypass combined with a subtotal or total gastrectomy, is performed routinely [24-28]. Published reports from these centers do not demonstrate increased complications.

Significance of this Study

Currently accepted surgical procedures all have significant long-term failure rates or frequently result in substantial malnutrition. Multiple new and novel surgical procedures are currently being tried that focus either on simple restriction or on increasing malabsorption. These new procedures are not designed with the intention of providing increased, permanent support for the patient's behavioral changes which are so critical in the long-term success of all bariatric surgery. The S.L.I.M.M.S. procedure is designed with the primary goal of a more sustained appetite suppression and increased early satiety.

Aims of This Study

The specific aim of the study is to assess the safety and efficacy of the S.L.I.M.M.S. Procedure as a stand-alone, single-stage bariatric operation.

METHODS

Trial Protocol

1. Patient Recruitment

   a. Recruitment into the study will be achieved by a physician awareness campaign using direct mail. An Internet awareness campaign will target potential patients. Announcements will include description of planned procedure, aim of study and experimental nature of the S.L.I.M.M.S. Procedure.
2. Patient Education

   a. Patient Education consisting of i. Detailed Consultation ii. Patient Education Packet iii. Written Examination iv. Education on pre- and post-operative dietary protocols v. Mandatory Dietary Rebuild counselling program vi. Permanent Surgical Weight Loss book provided vii. DietaryRebuild™ book provided viii. Exercise Instructions ix. Nutrition Supplementation Instructions
3. Patient Enrolment

   a. Enrolment into the study will be proceeded by patient education including a detailed discussion of the nature of this clinical trial. A detailed consent will also be provided.
4. Pre-trial Assessment

   1. Initial clinical assessment will include a detailed dietary history and a review for co-morbidities of obesity.
   2. Assessment of nutrition knowledge and quality of life will be obtained using the General Nutrition Knowledge Questionnaire, the Bariatric Quality of Life Index and the SF-36/Rand.
   3. Clinical assessment will include various weight parameters and measurement of serum glucose, hemoglobin A1c, lipids, vitamin levels, iron, ferritin, RBC folate, complete blood count, comprehensive metabolic profile, and abdominal ultrasound.
5. Surgery: S.L.I.M.M.S. Procedure
6. Patient Support

   1. In-clinic follow up
   2. Support groups offered
   3. Telephone-based group counselling sessions
7. Post-operative Assessment

   1. Weight Parameters measured at 6 months, 12 months and annually
   2. Laboratory assessment will include serum glucose, hemoglobin A1c, lipids, vitamin levels, iron, ferritin, RBC folate, complete blood count, comprehensive metabolic profile and lipid profile at 6 months, 12 months and annually thereafter
   3. Quality of life measure at 1, 12 and 24 months; Bariatric Quality of Life Index and SF-36/Rand

ELIGIBILITY:
Inclusion Criteria:

1. Be between 18 and 65 years of age
2. Have a body mass index of equal to or above 35 kgs per m2
3. Have identifiable obesity-related comorbidity; medical, physical or psycho-social
4. A history of attempts at weight reduction within the past five-year period
5. Ability to understand the non-surgical and surgical options for weight loss
6. Understand the behavioral changes needed to maximize surgical weight loss success
7. Agree to comply with recommended follow-up clinical assessments
8. Agree to comply with lifelong nutritional supplementation

Exclusion Criteria:

1. Lack of ability to understand weight loss options and requirements for long-term success with surgery
2. Inability to understand and accept the risks and potential benefits
3. Inability to understand and agree to the compliance requirements of the study
4. Prior gastric surgery including all forms of bariatric surgical or endoscopic procedures
5. A history of previous abdominal surgery which precludes gastric bypass
6. Medical contra-indications to bariatric surgery
7. Dementia, active psychosis, unstable psychiatric disease
8. Concurrent experimental drug use
9. Pregnancy or intending to conceive within 12 months or current breast-feeding
10. Recreational drug use or excessive alcohol intake
11. Use of drugs known to affect body composition
12. Use of cytotoxic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-10-26 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 6 months, 12 months and 2 years
  Primary efficacy variable is Weight Loss
  Weight loss will be measured as:
  1. Pounds lost (pre-op weight - post-op weight)
  2. Total Weight Loss, calculated as (Pre-op Weight-Current Weight) in pounds (lb)
  3. Percent Excess Weight Loss, calculated as [(Pre-op Weight - Ideal Body Weight)/Ideal Body Weight] x 100. Ideal Body Weight calculated using the universal IBW formula.

SECONDARY OUTCOMES:
Metabolic Comorbidity | 2 Years
  Glycemic control will be a specifically targeted endpoint. Serum glucose, HbA1c and documenting current diabetic medication regimen.
Changes in Quality of Life from baseline | 2 Years
  Quality of life measured using Bariatric Quality of Life Index and SF-36/Rand
Adverse Events | 2 Years
  Surgical complications are reported by participants and observed by the investigator and clinical trial staff, then reported on appropriate adverse event tracking forms

CONTACTS AND LOCATIONS:
Overall Officials: BRIAN QUEBBEMANN, M.D., Principal Investigator — The N.E.W. Program, Inc.
Locations (2):
- United States (2):
  - The N.E.W. Program, Inc., Newport Beach, California
  - Foothill Regional Medical Center, Tustin, California

IPD SHARING:
Plan to Share IPD: No